CLINICAL TRIAL: NCT06571409
Title: Clinical Evaluation of the Efficacy of a Dietary Supplement Claiming Anti-aging Properties and UV-protection in Healthy Adults: a Randomized, Double-blind, Placebo Controlled, Parallel, Clinical Trial
Brief Title: Clinical Evaluation of the Efficacy of a Dietary Supplement Claiming Anti-aging Properties and UV-protection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seppic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IT0003160/24
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Coriander Seed Oil - Dose 1 (Experimental): Dietary supplement - Coriander Seed Oil dose 1
  Interventions: Dietary Supplement: Coriander Seed Oil - Dose 1
- Coriander Seed Oil - Dose 2 (Experimental): Dietary supplement - Coriander Seed Oil dose 2
  Interventions: Dietary Supplement: Coriander Seed Oil - Dose 2
- Placebo (Placebo Comparator): Dietary supplement - Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Coriander Seed Oil - Dose 1 — The study foresees the intake of 1 capsule per day during 56 days
  Arms: Coriander Seed Oil - Dose 1
Dietary Supplement: Coriander Seed Oil - Dose 2 — The study foresees the intake of 1 capsule per day during 56 days
  Arms: Coriander Seed Oil - Dose 2
Dietary Supplement: Placebo — The study foresees the intake of 1 capsule per day during 56 days
  Arms: Placebo

SUMMARY:
The study aims to assess the anti-aging and photoprotective efficacy of two active concentrations of a food supplement composed of Coriander Seed Oil (CSO).

DETAILED DESCRIPTION:
A double blind, parallel groups, placebo-controlled study is carried out on 90 female subjects aged between 35 and 65 years old with visible Crow's feet wrinkles and mild to moderate skin slackness.

The study foresees 56 days of products intake. Evaluations of the parameters under study are performed at baseline, after 14, 28 and 56 days of products consumption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects
* Caucasian ethnicity
* Age between 35 and 65 years old (extremes included)
* Phototype I to III (with all skin types without any specific repartition)
* Visible Crow's feet wrinkles (> 2 according to Skin Aging Atlas - Caucasian Type - Bazin Roland) and mild to moderate skin slackness at cheek level (grade 1-3 - internal clinical scale)
* Subjects who have not been recently involved in any other similar study (at least 1 month of wash-out)
* Subjects registered with health social security or health social insurance
* Subjects having signed the Informed Consent Form (ICF) and Privacy Policy for their participation in the study and a photograph authorization
* Subjects able to understand the language used in the investigation center and the information given
* Subjects able to comply with the protocol and follow protocol constraints and specific requirements
* Willingness to use during all the study period only the product to be tested
* Willingness not to use similar products that could interfere with the expected product effect to be tested (e.g. with antiaging or soothing or UV protection efficacy)
* Willingness to not vary the normal daily routine (i.e. lifestyle, physical activity, diet etc.)
* Subjects under effective contraception (oral/not oral) if women of childbearing potential; not expected to be changed during the trial
* Subjects who have not sun exposure (both natural or artificial) for at least two months
* Subjects who accept not to expose in intensive way to UV rays during the whole study duration
* Subjects who have not been involved in any sun test (for SPF evaluation) or tests that provide skin irradiation since less than two months

Exclusion Criteria:

* Subject is taking part or planning to participate to another clinical study in the same or in another investigation center
* Subject who is deprived of freedom by administrative or legal decision or under guardianship
* Subject admitted in a sanitary or social facilities
* Subject who is planning an hospitalization during the study
* Subjects under treatment with food supplements which could interfere with the functionality of the product under study
* Subject breastfeeding, pregnant or not willing to take necessary precautions to avoid pregnancy during the study (if women of childbearing potential)
* Subject has started or changed estrogen-progesterone contraception or hormonal treatment, within the 3 months prior to the study or foreseeing it for the duration of the study
* Subject having an acute, chronic or progressive illness liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
* Subjects under radiotherapy, chemotherapy at any time
* Subject having a skin condition liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
* Pharmacological treatments (topic or systemic) known to interfere with skin metabolism/physiology
* Subjects under locally pharmacological/non-pharmacological treatment applied on the skin area monitored during the test
* Subject with known or suspected sensitization to one or more test formulation ingredients
* Subjects considered as not adequate to participate to the study by the investigator
* Adult protected by law (under control or hospitalized in public or private institutions for reasons other than research, or incarcerated)
* Subjects not able to communicate or cooperate with the investigator for problems related to language, mental retardation or impaired brain function

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Skin profilometry | Baseline
  Primos 3D
Skin profilometry | 14 days
  Primos 3D
Skin profilometry | 28 days
  Primos 3D
Skin profilometry | 56 days
  Primos 3D

SECONDARY OUTCOMES:
Skin elasticity | Baseline
  Cutometer
Skin elasticity | 14 days
  Cutometer
Skin elasticity | 28 days
  Cutometer
Skin elasticity | 56 days
  Cutometer
Transepidermal water loss | Baseline
  Tewameter
Transepidermal water loss | 14 days
  Tewameter
Transepidermal water loss | 28 days
  Tewameter
Transepidermal water loss | 56 days
  Tewameter
Erythema index | Baseline
  Skin haemoglobin quantification by Mexameter 24h after UV exposure
Erythema index | 28 days
  Skin haemoglobin quantification by Mexameter 24h after UV exposure
Erythema index | 56 days
  Skin haemoglobin quantification by Mexameter 24h after UV exposure
Skin inflammation (subgroup of 20 subjects) | Baseline
  TNF-alpha quantification by Enzyme-Linked Immunosorbent Assay on skin stripping performed before and 24h after UV exposure
Skin inflammation (subgroup of 20 subjects) | 56 days
  TNF-alpha quantification by Enzyme-Linked Immunosorbent Assay on skin stripping performed before and 24h after UV exposure
Skin lipoxidation (subgroup of 20 subjects) | Baseline
  Malondialdehyde quantification by spectrophotometry on skin stripping performed before and 4h and 24h after UV exposure
Skin lipoxidation (subgroup of 20 subjects) | 56 days
  Malondialdehyde quantification by spectrophotometry on skin stripping performed before and 4h and 24h after UV exposure
Self-assessment of product efficacy | 56 days
  Questionnaire (10 questions with 4 possible answers : completely agree / agree / disagree / completely disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Spartà, Study Director — Complife Italia S.r.l
Locations (1):
- Complife Italia S.r.l, San Martino Siccomario, Italy

IPD SHARING:
Plan to Share IPD: No